CLINICAL TRIAL: NCT03665389
Title: Evaluation of Fractional Flow Reserve Calculated by Computed Tomography Coronary Angiography in Patients Undergoing Transcatheter Aortic Valve Replacement（FORTUNA）: Single Center, Open-label, Exploratory, Prospective Study
Brief Title: Evaluation of Fractional Flow Reserve Calculated by Computed Tomography Coronary Angiography in Patients Undergoing TAVR
Acronym: FORTUNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kobe University (Industry)
Responsible Party: Principal Investigator, Hiromasa Otake, Senior Lecturer, Kobe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 300028
Record Dates: First submitted 2018-08-30; First posted 2018-09-11 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Aortic Valve Stenosis; Coronary Artery Disease
Keywords: FFRct; aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Among patients who undergo TAVR at the kobe university hospital, those who are found to have moderate or severe stenosis on cCTA performed before surgery and judged to clinically require ischemia evaluation will be included in this study.
  Interventions: Device: iFR / FFR measurement

INTERVENTIONS:
Device: iFR / FFR measurement — At the time of pre-TAVR coronary angiogram, iFR (iFR before TAVR) will be measured. The cCTA data collected from patients whose consent is obtained following TAVR will be anonymized and sent to HeartFlow, Inc., where the FFRct （FFRct before TAVR） values will be calculated using their cardiovascular dynamics analysis program. With the FFRct values blinded, FFR (FFR after TAVR) and iFR (iFR after TAVR) will be measured using a guide wire that is capable of sensing pressure after TAVR is performed. Furthermore, FFRct(FFRct after TAVR) is calculated from cCTA taken after TAVR.

SUMMARY:
The objective of this study is to evaluate the relationship between fractional flow reserve (FFR) derived from coronary computed tomography angiography (FFRct) before transcatheter aortic valve replacement (TAVR) and FFR after TAVR so as to investigate whether FFRct is useful for evaluating myocardial ischemia of severe AS. Furthermore, by measuring the instantaneous wave-free ratio (iFR) which is a physiological diagnostic method of coronary artery stenosis before and after TAVR and comparing iFR (iFR before and after TAVR) and FFR (FFR after TAVR) with FFRct (FFRct before and after TAVR), It also aims to deepen understanding of resting coronary artery physiology in aortic valve stenosis.

DETAILED DESCRIPTION:
This is a single-center, open-label, exploratory, prospective study. Among patients who undergo coronary computed tomography angiography (cCTA) prior to TAVR, those with moderate or severe stenotic lesions will be included in the study. Patients from whom consent is obtained following TAVR will be enrolled in the study.

Among patients who undergo TAVR at the Kobe University Hospital from September 2018 to March 2022, those who are found to have moderate or severe stenosis on cCTA performed before surgery and judged to clinically require ischemia evaluation will be included in the study. At the time of pre-TAVR coronary angiogram, iFR (iFR before TAVR) will be measured. The cCTA data collected from patients whose consent is obtained following TAVR will be anonymized and sent to HeartFlow, Inc., where the FFRct（FFRct before TAVR) values will be calculated using their cardiovascular dynamics analysis program. FFR (FFR after TAVR) and iFR (iFR after TAVR) will be measured using a guide wire that is capable of sensing pressure after TAVR is performed. Furthermore, FFRct (FFRct after TAVR) is calculated from cCTA taken after TAVR.

ELIGIBILITY:
Inclusion Criteria:

1. Among patients who have undergone cCTA prior to TAVR, those with moderate stenotic lesions (30 to <70%) or severe stenotic lesions on CT who are candidates for percutaneous coronary intervention (PCI) following TAVR
2. Patients aged 20 years or older at the time of diagnosis

Exclusion Criteria:

Patients who meet any one of the following criteria will be excluded from this study:

1. Patients who were implanted with metal stents in the left main trunk,
2. Patients with stenosis of >30% in the left main trunk who were implanted with at least one metal stent in the vessel(s) of the left coronary circulation,
3. Patients who were implanted with metal stents in at least 2 vessels of the coronary circulation,
4. Patients who requested withdrawal of consent for participation in this research study after providing their consent,
5. Patients who underwent coronary artery bypass surgery,
6. Patients with coronary artery chronic total occlusion,
7. Patients who developed acute myocardial infarction in the past 2 months,
8. Patients whose cCTA was determined to be unreadable during its evaluation at the study site because of the presence of artifacts which were severe enough to cause problems with the angiogram,
9. Patients who were judged by the principal investigator to be unsuitable for the study for other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-09-13 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
FFRct before TAVR | Baseline

SECONDARY OUTCOMES:
FFRct after TAVR | Up to 4 weeks
FFR after TAVR | Up to 4 weeks
iFR before TAVR and after TAVR | Baseline and up to 4 weeks
Stenosis degree in coronary angiography performed before TAVR | Baseline